CLINICAL TRIAL: NCT04937985
Title: Validity and Test-Retest Reliability of Unsupported Upper Limb Exercise Test in Patients With Chronic Neck Pain
Brief Title: Unsupported Upper Extremity Exercise Test in Chronic Neck Pain
Status: Completed | Type: Observational
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Ilknur Naz, Assoc. Prof, Izmir Katip Celebi University
Other Study IDs: IKC3
Record Dates: First submitted 2021-06-18; First posted 2021-06-24 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Neck Pain; Upper Extremity Dysfunction
Keywords: chronic neck pain; upper extremity test; validity; reliability
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- UULEX Test Group: Patients with chronic neck pain
  Interventions: Other: Performance Tests

INTERVENTIONS:
Other: Performance Tests — Performance tests consist of Six Minute Pegboard Ring Test, 30-Second Push-Up Test and Arm, Shoulder and Hand Injury Questionnaire (DASH), Neck Disability Index, New York Posture Rating Chart and Short Form-36 Health Survey.

SUMMARY:
The aim of this study was to examine the validity and test-retest reliability of unsupported upper extremity exercise test (UULEX) in individuals with chronic neck pain.

Patients with neck pain lasting at least 3 months will be included in the study. It is planned to examine the validity and test-retest reliability of the UULEX test in that patient groups.

DETAILED DESCRIPTION:
Persons with chronic neck pain may limit the functional use of their upper extremities. It is recommended to determine appropriate upper extremity measurement methods in patients with chronic neck pain. Therefore the aim of this study was to examine the validity and test-retest reliability of unsupported upper extremity exercise test (UULEX) in individuals with chronic neck pain.

Six Minute Pegboard Ring Test, 30-Second Push-Up Test and Arm, Shoulder and Hand Injury Questionnaire (DASH), Visual Analog Scale, Neck Disability Index, New York Posture Rating Chart and Short Form-36 Health Survey were used to evaluate the validity of the test. For test-retest reliability, the unsupported upper extremity test was repeated 1 week later by the same investigator.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old

Exclusion Criteria:

* Presence of additional disease affecting upper extremity and hand functions (carpal tunnel syndrome, trigger finger, impingement syndrome,thoracic outlet syndrome, lateral and medial epicondylitis, hand osteoarthritis, etc.),
* having undergone upper extremity or cervical region surgery
* cervical radiculopathy, rheumatic disease, presence of neurological symptoms
* According to the Visual Analogue Scale (VAS), neck pain intensity in activity is less than 3,
* Acute or chronic respiratory illness
* Cardiac disease
* Problem recognizing verbal commands
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 44 patients with neck pain lasting at least 3 months and being volunteer to participate in our study
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Functional capacity test | 15 minutes- Change from baseline values at 1 week
  Unsupported Upper Limb Exercise Test

SECONDARY OUTCOMES:
Functional capacity test | 6 minutes (single application)
  Six minute pegboard ring test
Upper extremity endurance test | 30 seconds (single application)
  30 Second Push Up Test
Disability Level | 15 minutes (single application)
  Neck Disability Index: Scores range from 0 to 50, with higher scores indicating higher disability
Upper Extremity Function | 15 minutes (single application)
  Disability of Arm Shoulder and Hand Injury Questionnaire: Scores range from 0 to 100, with higher scores indicating higher disability
Severity of Pain | 3 minutes (single application)
  Visual analog Scale:Scores range from 0 to 100, with higher scores indicating higher pain severity
Postural Assessment | 10 minutes (single application)
  New York Posture Rating Chart :Scores range from 13 to 65, with higher scores indicating better posture
Quality of Life Assessment | 15 minutes
  Short Form-30 Health Survey: Scores range from 0 to 100, with higher scores indicating better quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Karazeybek, Principal Investigator — Izmir Katip Celebi University; İlknur Naz, Study Director — Izmir Katip Celebi University
Locations (1):
- İlknur Naz Gürşan, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No